CLINICAL TRIAL: NCT03184675
Title: Main Researcher for the Effects of Functional Action-observation Training on Gait Ability
Brief Title: The Effects of Functional Action-Observation Training on Gait Ability in Patients With Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Do hyun Kim, primary researcher, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: InjeU 2
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional action observation training (Experimental)
  Interventions: Other: Functional action observation training
- General action observation training group (Other)
  Interventions: Other: General action observation training

INTERVENTIONS:
Other: Functional action observation training — the Four Square Step Test (FSST) performance video for enhancing the dynamic balance and the video including participants' daily activities to increase the gait ability such as walking in a corridor, walking around the hospital, walking to the therapy room, coming out of the ward after opening and closing the door of it, coming in and out of toilet, shifting their blue plate. and bringing something from a refrigerator were produced and watched.
  Arms: Functional action observation training
Other: General action observation training — step 1, looking at the front, while walking comfortably; step 2, looking left and right, while walking; step 3, looking up and down, while walking; step 4, looking at the front, left and right, up and down while walking. After 15 minutes of watching the video, the exercise program with a therapist was conducted to increase the gait ability, for 15 minutes.
  Arms: General action observation training group

SUMMARY:
This study aimed to examine the effects of functional action observation training on gait ability in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis with stroke through computed tomography or magnetic resonance imaging, more than six months ago.
2. determination not to have cognitive disability, based on the score(>24 point) of mini mental state examination-Korea version.
3. determination not to have visual abnormalities including the unilateral neglect through the motor-free visual perception test(MVPT)
4. ability to independently gait longer than 10m in the room and to keep standing up without help.

Exclusion Criteria:

1. surgery in the last three months
2. participating any other research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2017-07-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
temporal gait variables | 8 weeks
  gait velocity